CLINICAL TRIAL: NCT01970813
Title: Efficacy of Acupuncture and Bee Venom Acupuncture on Patients With Idiopathic Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kyunghee University Medical Center (Other)
Responsible Party: Principal Investigator, Seong-Uk Park, Associate professor, Kyunghee University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NRF-2011-0021389
Record Dates: First submitted 2013-10-17; First posted 2013-10-28 (Estimated); Last update posted 2015-09-09 (Estimated); Status verified 2015-09

CONDITIONS: Idiopathic Parkinson's Disease
Keywords: Parkinson's disease; Idiopathic Parkinson's disease; acupuncture; bee venom acupuncture
MeSH Terms: conditions — Parkinson Disease | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Study group (Active Comparator): acupuncture and bee venom acupuncture point injection
  Interventions: Device: acupuncture and bee venom acupuncture point injection
- Control group (Sham Comparator): sham acupuncture and normal saline injections
  Interventions: Device: sham acupuncture and normal saline injections
- Waiting group (No Intervention): no additional intervention

INTERVENTIONS:
Device: acupuncture and bee venom acupuncture point injection — acupuncture and bee venom acupuncture point injection at 10 acupuncture points twice a week for 12 weeks. This intervention is added on to the conventional antiparkinsonian drugs.
  Arms: Study group
Device: sham acupuncture and normal saline injections — sham acupuncture and normal saline injections at 10 sham acupuncture points twice a week for 12 weeks. This intervention is added on to the conventional antiparkinsonian drugs.
  Arms: Control group

SUMMARY:
The aim of this study is to evaluate the efficacy of acupuncture and bee venom acupuncture (BVA) for idiopathic Parkinson's disease (IPD) through a sham-controlled trial and investigate whether there is sustainability of treatments effects by follow-up assessments after the end of the treatment.

DETAILED DESCRIPTION:
A total of 90 patients with idiopathic Parkinson's disease (IPD) who have been on a stable dose of anti-parkinsonian medication for at least one month with two or more symptoms among tremor, rigidity, postural instability, and bradykinesia will be included in this study. Participants will be randomly assigned to the study, the control, or the waiting group (2:2:1).

Initial assessment will be performed with the Unified Parkinson's Disease Rating Scale (UPDRS) parts II and III, the Parkinson's Disease Quality of Life Questionnaire (PDQL), the Beck Depression Inventory (BDI), and evaluation of the 20-m walking time and the steps to walk 20-m, as well as postural instability.

Acupuncture and BVA treatments will then be performed on the study group, and sham acupuncture and normal saline injections will be performed on the control group twice a week for 12 weeks. The waiting group does not receive any added treatment during the 12 weeks.

The initial assessment will be repeated after 12 weeks in all groups. In the study and the control groups, an additional assessment will be repeated after 16 and 20 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients with IPD who have been on a stable dose of anti-parkinsonian medication for at least one month.
* Hoehn & Yahr scale I-IV
* More than one point in two or more items (tremor, rigidity, postural instability, and bradykinesia) in the UPDRS Part III, etc.

Exclusion Criteria:

* Severe psychiatric or organic brain disorders other than PD, previous or current
* Secondary Parkinsonism due to cerebrovascular disease, tumor, infection, etc.
* Atypical Parkinsonian or Parkinson plus syndrome

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2012-10; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Change of the Unified Parkinson's Disease Rating Scale (UPDRS) parts II and III | baseline, up to 12 weeks, 16 weeks, and 20 weeks
  The UPDRS part II is evaluation of the activities of daily living (ADL) and part III is the motor examination.

CONTACTS AND LOCATIONS:
Overall Officials: Seong-Uk Park, Ph.D, Principal Investigator — Kyunghee University
Locations (1):
- Kyung Hee University Hospital at Gangdong, Seoul, South Korea